CLINICAL TRIAL: NCT01854554
Title: A Prospective Phase II Randomized Trial to Compare Intensity Modulated Proton Radiotherapy (IMPT) vs. Intensity Modulated Radiotherapy (IMRT) for Newly Diagnosed Glioblastoma (WHO Grade IV)
Brief Title: Glioblastoma Multiforme (GBM) Proton vs. Intensity Modulated Radiotherapy (IMRT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0097; NCI-2013-01089 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Results first posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Brain Cancer
Keywords: Brain cancer; Glioblastoma; Glioblastoma Multiforme; GBM; Intensity Modulated Proton Radiotherapy; IMPT; Intensity Modulated Radiotherapy; IMRT; Radiotherapy; XRT; Cognitive tests; Thinking skills tests; Questionnaires; Surveys; Quality of life; QOL
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma | interventions — Radiotherapy; Neuropsychological Tests; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intensity Modulated Proton Radiotherapy (IMPT) (Experimental): IMPT treatments delivered as once daily fractions, 5 days per week Monday - Friday for 30 treatments.
  Interventions: Radiation: IMPT; Behavioral: Cognitive Tests; Behavioral: Questionnaires
- Intensity Modulated Radiotherapy (IMRT) (Experimental): IMRT treatments delivered as once daily fractions, 5 days per week Monday - Friday for 30 treatments.
  Interventions: Radiation: IMRT; Behavioral: Cognitive Tests; Behavioral: Questionnaires

INTERVENTIONS:
Radiation: IMPT — IMPT treatments delivered as once daily fractions, 5 days per week Monday - Friday for 30 treatments.
  Other Names: Radiotherapy; XRT
  Arms: Intensity Modulated Proton Radiotherapy (IMPT)
Radiation: IMRT — IMRT treatments delivered as once daily fractions, 5 days per week Monday - Friday for 30 treatments.
  Other Names: Radiotherapy; XRT
  Arms: Intensity Modulated Radiotherapy (IMRT)
Behavioral: Cognitive Tests — Cognitive tests given at baseline, 4 months, then every 2 months for 2 years.
  Other Names: Thinking skills tests
Behavioral: Questionnaires — Questionnaires about quality of life and symptoms given at baseline, 4 months, then every 2 months for 2 years.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to compare IMRT with IMPT in patients with glioblastoma. Researchers want to learn about cognitive side effects (mental status changes) that may occur, such as memory loss and impaired thinking.

IMRT is the delivery of focused radiation therapy using photon beams and advanced computer planning to help shape the dose in order to give the highest possible dose to the tumor with the least dose to surrounding normal tissues.

IMPT is also focused radiation therapy similar to IMRT, but it uses proton particles to deliver the radiation instead of photon beams. IMPT also uses advanced computer planning in order to shape the dose to the target with the least dose to surrounding normal tissues.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. You will have an equal chance of being assigned to either group.

If you are in Group 1, you will receive IMRT.

If you are in Group 2, you will receive IMPT.

Radiation Therapy:

In both groups, you will receive radiation treatments each day, Monday-Friday, starting on Day 1. You will continue to receive radiation treatment until you have completed 30 total treatments. This is a total of up to 6 weeks of treatment.

You will sign a separate consent form for the IMRT or IMPT that will explain the procedures and risks in detail.

Study Visits:

Before beginning radiation, you will have what is called a "simulation" to plan your radiation. During the simulation, you will be flat on your back on a computed tomography (CT) table and a soft plastic mask will be made to help hold your head still during treatment. This is the position you will be in when you receive radiation treatment. You will then have a CT scan, which will make computerized images to help plan your treatment.

At Month 2 (+/- 30 days):

* You will have a physical exam, including measurement of your vital signs.
* You will have an MRI to check the status of the disease.
* You will be asked about any drugs you may be taking and side effects you may be having.
* You will complete the thinking skills tests and the questionnaires about your quality of life and symptoms.

Length of Treatment:

You may receive up to 6 weeks of radiation therapy. You will no longer be able to receive radiation therapy if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your active participation on the study will be over after the follow-up visits.

Follow-Up:

At Month 4 (+/- 30 days) and then every 2 months for up to 2 years after radiation therapy:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any side effects you may be having.
* You will have an MRI to check the status of the disease.
* You will complete the thinking skills tests and the questionnaires about your quality of life and symptoms.

Starting 2 years after radiation therapy, the study staff will continue checking your medical record to find out about your health status from then on.

This is an investigational study. IMRT is delivered using FDA-approved and commercially available methods. IMPT is investigational.

Up to 90 participants will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of: Glioblastoma or Gliosarcoma (WHO Grade IV) adapted RPA class III, IV, or V.
2. All patients must be >/=18 years of age.
3. All patients must sign informed consent verifying that they are aware of the investigational nature of this study in keeping with the rules and policies of MD Anderson Cancer Center. The only acceptable consent form is the one approved by MD Anderson IRB.
4. All patients must have a baseline Mini Mental Status Examination score >/=21.
5. All patients must have a KPS >/=70.
6. All patients must be eligible to have either IMRT or IMPT as determined by the study radiation oncologist.
7. All patients must be able to undergo MRI with and without contrast with a glomerular filtration rate (eGFR) greater than or equal to 30 mg/min/1.72 m2.
8. All patients must have adequate liver, renal, and hematologic function within 14 days of registration as defined by Aspartate Amino Transferase (AST)/Alanine Amino Transferase (ALT)/Alkaline Phosphatase < 3 times normal, creatinine </=1.7 mg/dl, BUN </= 35mg/dl, absolute neutrophil count >/=1,800 cells/mm3, Hemoglobin >/= 10 g/dl, and platelet count > 100,000.
9. All patients must be able to adequately read, write and speak to participate in the cognitive and quality of life assessments. However mild to moderate deficits in these functions due to tumor are allowed.

Exclusion Criteria:

1. Patients will be excluded if they are not planning to receive concurrent temozolomide.
2. Patients will be excluded if they have had prior radiation to the brain.
3. Patients will be excluded if they have had prior surgical resection of brain for other brain tumors.
4. Patients will be excluded if they are pregnant as assessed by serum beta human chorionic gonadotropin (b-HCG). A serum b-HCG test will be performed no greater than 14 days prior to study registration for women of childbearing potential.
5. Patients with gliomatosis will be excluded.
6. Patients with Gliadel bis-chloroethylnitrosourea (BCNU) implanted wafers will be excluded.
7. Patients weighing greater than 136 kilograms will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-05-17 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Chung, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Details: May 2013- March 2016. All participants recruited at UT MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Intensity Modulated Proton Radiotherapy (IMPT) | Intensity Modulated Radiotherapy (IMRT)
Started | 42 | 48
Completed | 28 | 39
Not Completed | 14 | 9
Not completed — Denial of Insurance Coverage | 12 | 0
Not completed — Decided to get treatment locally | 1 | 5
Not completed — Received IMR only due to insurance analysis | 1 | 0
Not completed — Did Not Meet Eligibility Criteria | 0 | 2
Not completed — Progression | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Between June 2013 and March 2016, 90 patients consented to participate and 67 were treated (28 PT, 39 IMRT) with the majority of patients excluded before treatment began due to insurance denial of proton therapy
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensity Modulated Proton Radiotherapy (IMPT) | Intensity Modulated Radiotherapy (IMRT) | Total
Number analyzed (Participants) | 28 | 39 | 67
Age, Continuous [Median (Full Range); unit: years] | 53 [26 to 82] | 55 [33 to 72] | 53.8 [26 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 19 | 31
  Male | 16 | 20 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26 | 31 | 57
  Hispanic | 1 | 5 | 6
  African American | 1 | 2 | 3
  Asian | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 39 | 67

OUTCOME MEASURES:

1. Primary Outcome: Time to Cognitive Failure
Description: Time to cognitive failure on any of 6 primary variables from pre-specified cognitive tests (HVLT-R total recall, HVLT-R delayed recall, HVLT-R delayed recognition, TMT Part A or Part B, COWA) with failure defined as a decline that meets or exceeds the reliable change index (RCI) for each cognitive test variable. A cumulative incidence approach used to estimate median time to cognitive failure in order to account for the competing risks of disease progression and death.
Time Frame: baseline, 4 months, then every 2 months for 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Intensity Modulated Radiotherapy (IMRT) | Intensity Modulated Proton Radiotherapy (IMPT)
Number analyzed (Participants) | 35 | 24
months | 7.7 [4.2 to NA] — Not estimable | 4.9 [3.3 to NA] — Not estimable
Statistical Analysis 1: Comparison: Intensity Modulated Radiotherapy (IMRT) vs Intensity Modulated Proton Radiotherapy (IMPT); Test type: Superiority; p = .74, Gray's test; Cumulative Incidence Function treating progressive disease (RANO) or death before cognitive function decline as a competing risk

2. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as time from registration/randomization to the date of death from any cause. Overall survival rates are estimated by the Kaplan-Meier method.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Population: Between June 2013 and March 2016, 90 participants consented to participate and 67 (41 and 26 participants effectively treated with IMRT and IMPT) were treated with the majority of participants excluded before treatment began due to insurance denial of proton therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Intensity Modulated Radiotherapy (IMRT) | Intensity Modulated Proton Radiotherapy (IMPT)
Number analyzed (Participants) | 41 | 26
months | 21.2 [16.4 to 33.7] | 24.5 [17.3 to 34.8]
Statistical Analysis 1: Comparison: Intensity Modulated Radiotherapy (IMRT) vs Intensity Modulated Proton Radiotherapy (IMPT); Test type: Superiority; p = .60, Log Rank

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Measured from date of registration to date of first observation of progressive disease, symptomatic deterioration or death due to any cause. Participants last known to be alive and progression-free are censored at date of last contact.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
Population: Between June 2013 and March 2016, 90 patients consented to participate and 67 (41 and 26 participants effectively treated with IMRT and IMPT) were treated with the majority of participants excluded before treatment began due to insurance denial of proton therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Intensity Modulated Radiotherapy (IMRT) | Intensity Modulated Proton Radiotherapy (IMPT)
Number analyzed (Participants) | 41 | 26
months | 8.9 [7.6 to 13.6] | 6.6 [3.9 to 14.3]
Statistical Analysis 1: Comparison: Intensity Modulated Radiotherapy (IMRT) vs Intensity Modulated Proton Radiotherapy (IMPT); Test type: Superiority; p = 0.24, Log Rank

4. Secondary Outcome: Number of Participants Experienced Adverse Events by Maximum Grade (Grade 2 or Higher)
Description: The adverse severity was graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v4.0).
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL
  Grade 4 Life-threatening consequences; urgent intervention indicated.
  Count of participants experiencing adverse events. Should a participant experience multiple adverse events at different grades, the patient is counted only once at the highest grade.
Time Frame: 2 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Intensity Modulated Radiotherapy (IMRT) | Intensity Modulated Proton Radiotherapy (IMPT)
Number analyzed (Participants) | 41 | 26
Participants
  Grade 4 Adverse Events | 2 | 1
  Grade 3 Adverse Events | 4 | 2
  Grade 2 Adverse Events | 14 | 5

ADVERSE EVENTS:
Time Frame: 2 years
Description: During this study, both the Intensity Modulated Radiotherapy (IMRT) and Intensity Modulated Proton Radiotherapy (IMPT) arms reported serious and life-threatening adverse events. Specifically, 2 participants in the IMRT arm and 1 participant in the IMPT arm experienced Grade 4 life-threatening events that required urgent intervention
Arm/Group | Intensity Modulated Radiotherapy (IMRT) | Intensity Modulated Proton Radiotherapy (IMPT)
All-Cause Mortality (participants affected / at risk) | 29/41 | 22/26
Serious Adverse Events (participants affected / at risk) | 2/41 | 1/26
Other Adverse Events (participants affected / at risk) | 29/41 | 19/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intensity Modulated Radiotherapy (IMRT) (N=41) | Intensity Modulated Proton Radiotherapy (IMPT) (N=26)
Platelet count decreased (Blood and lymphatic system disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intensity Modulated Radiotherapy (IMRT) (N=41) | Intensity Modulated Proton Radiotherapy (IMPT) (N=26)
Alopecia (Skin and subcutaneous tissue disorders) | 29 | 19
Fatigue (General disorders) | 26 | 17
Headache (Nervous system disorders) | 20 | 8
Agitation (Psychiatric disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 9 | 4
Anxiety (Nervous system disorders) | 3 | 1
Ataxia (Nervous system disorders) | 3 | 1
Blurred vision (Eye disorders) | 1 | 1
Confusion (Psychiatric disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 6 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Depression (Psychiatric disorders) | 2 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 17 | 18
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 7 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 3
Dysarthria (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphasia (Nervous system disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 | 0
Edema face (General disorders) | 3 | 1
Edema limbs (General disorders) | 3 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 1
Facial nerve disorder (Nervous system disorders) | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gastroparesis (Gastrointestinal disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Hydrocephalus (Nervous system disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 6 | 5
Irritability (General disorders) | 1 | 0
Localized edema (General disorders) | 1 | 1
Malaise (General disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 2 | 3
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 15 | 4
Neck edema (General disorders) | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Nystagmus (Nervous system disorders) | 1 | 0
Olfactory nerve disorder (Nervous system disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 2
Pain (General disorders) | 1 | 1
Paresthesia (Nervous system disorders) | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Platelet count decreased (Investigations) | 4 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 1
Scrotal pain (Reproductive system and breast disorders) | 1 | 0
Seizure (Nervous system disorders) | 6 | 2
Sinus pain (Nervous system disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT01854554/Prot_SAP_000.pdf